CLINICAL TRIAL: NCT00110357
Title: Phase I Study of Erbitux™ (Cetuximab) in Pediatric Patients With Refractory Solid Tumors
Brief Title: Study of Erbitux™ (Cetuximab) in Pediatric Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CA225-085
Record Dates: First submitted 2005-05-06; First posted 2005-05-09 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Cancer; Refractory Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): 1-12 years old
  Interventions: Drug: Cetuximab + Irinotecan
- Group B (Active Comparator): 13-18 years old
  Interventions: Drug: Cetuximab + Irinotecan

INTERVENTIONS:
Drug: Cetuximab + Irinotecan — Intravenous (IV) cetuximab 75 - 250 mg/m2 depending on dose escalation for MTD, weekly; irinotecan was administered at a dose of 16 or 20 mg/m2 or per dose escalation, administered x5 days x2 weeks, separated by 2 days off, every 21 days.
  Arms: Group A
Drug: Cetuximab + Irinotecan — Intravenous (IV) cetuximab 75 - 250 mg/m2 depending on dose escalation for MTD, weekly; irinotecan was administered at a dose of 20 mg/m2 or per dose escalation, administered x5 days x2 weeks, separated by 2 days off, every 21 days.
  Arms: Group B

SUMMARY:
The purpose of this clinical research study is to establish the maximum tolerated dose and recommended Phase II dose of Erbitux™ in combination with Irinotecan in pediatric and adolescent patients with refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of a solid tumor which has progressed on, or following standard therapy, or for which no standard effective therapy is known.
* Children age 1-18 years.

Exclusion Criteria:

* Presence of active infection.
* Requirement to receive concurrent chemotherapy immunotherapy, radiotherapy, or any other investigational drug while on study.
* Inadequate bone marrow, hepatic, or renal function.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - University Of Arizona Health Sciences Center, Tucson, Arizona
  - The Children'S Hospital, Denver, Colorado
  - University Of Florida, Gainesville, Florida
  - Children'S Healthcare Of Atlanta, Atlanta, Georgia
  - Sidney Kimmel Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University Medical Center Infectious Diseases, Nashville, Tennessee
  - University Of Texas Md Anderson Cancer Ctr, Houston, Texas

REFERENCES:
- [Background] Trippett TM, Herzog C, Whitlock JA, Wolff J, Kuttesch J, Bagatell R, Hunger SP, Boklan J, Smith AA, Arceci RJ, Katzenstein HM, Harbison C, Zhou X, Lu H, Langer C, Weber M, Gore L. Phase I and pharmacokinetic study of cetuximab and irinotecan in children with refractory solid tumors: a study of the pediatric oncology experimental therapeutic investigators' consortium. J Clin Oncol. 2009 Oct 20;27(30):5102-8. doi: 10.1200/JCO.2008.20.8975. Epub 2009 Sep 21. PMID 19770383

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 48 subjects were enrolled; 1 additional subject withdrew informed consent before any measurements or treatment. 46 subjects (27 in the 1- to 12-yrs-old group and 19 subjects in the 13- to 18-yrs-old group) were treated; 2 subjects in the 13-18 yrs group were not treated, and are NOT included in Participant Flow or Baseline Characteristics tables.
Period: Overall Study
Arm/Group | 1- to 12-years-old | 13- to 18-years-old
Started | 27 | 19
Completed | 0 (Number Still on Study) | 0 (Number Still on Study)
Not Completed | 27 | 19
Not completed — Deterioration without progression | 2 | 0
Not completed — Disease progression/relapse | 20 | 15
Not completed — Study Closure | 1 | 0
Not completed — Study Drug Toxicity | 1 | 3
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1- to 12-years-old | 13- to 18-years-old | Total
Number analyzed (Participants) | 27 | 19 | 46
Age, Continuous [Median (Full Range); unit: years] | 8.0 [1.0 to 12.0] | 16.0 [13.0 to 18.0] | 10 [1.0 to 18.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 12 | 10 | 22
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 2 | 2
  Black or African American | 5 | 2 | 7
  White | 21 | 14 | 35
  Other | 1 | 1 | 2
Disease diagnosis [Number; unit: Participants]
  CNS Primary Tumor | 17 | 9 | 26
  Non-CNS Primary Tumor | 10 | 10 | 20
Performance Status [Number; unit: Participants] — For participants ≤10 years of age, Lansky play scale is used; for participants >10 years of age, Karnofsky scale is used. The Lansky scale runs from 100 to 0, where 100 is "fully active/normal" and 0 is "unresponsive." Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death.
  Participants
    >70-100 | 19 | 16 | 35
    ≥50-70 | 8 | 3 | 11
    <50 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With a Dose-Limiting Toxicity
Description: Dose-limiting toxicities (DLTs)=serious drug side effects preventing further dose escalation. If 1 of the first 3 subjects developed a DLT during cycle 1 up to 3 additional subjects were enrolled at that dose level. The maximum dose level at which DLTs occurred in fewer than 2 out of 3 to 6 subjects was defined as the Maximum Tolerated Dose (MTD).
Time Frame: Prior to each 21-day cycle until dose-limiting toxicities
Population: All treated subjects
Measure: Number; unit: Participants
Groups:
- Group A: 75/20: Cetuximab 75 mg/m2 + Irinotecan 20 mg/m2 in participants 1-12 years
- Group A: 150/20: Cetuximab 150 mg/m2 + Irinotecan 20 mg/m2 in participants 1-12 years of age
- Group A 150/16: Cetuximab 150 mg/m2 + Irinotecan 16 mg/m2 in participants 1-12 years of age
- Group A: 250/16: Cetuximab 250 mg/m2 + Irinotecan 16 mg/m2 in participants 1-12 years of age
- Group B: 75/20: Cetuximab 75 mg/m2 + Irinotecan 20 mg/m2 in participants 13-18 years of age
- Group B: 150/20: Cetuximab 150 mg/m2 + Irinotecan 20 mg/m2 in subjects 13-18 years of age
- Group B: 250/20: Cetuximab 250 mg/m2 + Irinotecan 20 mg/m2 in participants 13-18 years of age
Arm/Group | Group A: 75/20 | Group A: 150/20 | Group A 150/16 | Group A: 250/16 | Group B: 75/20 | Group B: 150/20 | Group B: 250/20
Number analyzed (Participants) | 6 | 6 | 3 | 12 | 8 | 4 | 7
Participants
  Subjects with a dose-limiting toxicity | 1 | 2 | 0 | 0 | 1 | 0 | 1
  Subjects with no dose-limiting toxicity | 5 | 4 | 3 | 12 | 7 | 4 | 6

2. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: The single dose pharmacokinetics (PK) of cetuximab was administered with an intravenous dose of irinotecan 16 to 20 mg/m2; Cmax was evaluated based on concentration-time profile.
Time Frame: up to 168 hours after the start of the cetuximab infusion during the first 21-day cycle of the study
Measure: Geometric Mean (Standard Deviation); unit: µg/mL
Groups:
- Group A: 75: Cetuximab 75 mg/m2 + Irinotecan 16-20 mg/m2 in participants 1-12 years
- Group A :150: Cetuximab 150 mg/m2 + 16-20 mg/m2 in participants 1-12 years of age
- Group A: 250: Cetuximab 250 mg/m2 + Irinotecan 16-20 mg/m2 in participants 1-12 years of age
- Group B: 75: Cetuximab 75 mg/m2 + Irinotecan 16-20 mg/m2 in participants 13-18 years of age
- Group B: 150: Cetuximab 150 mg/m2 + Irinotecan 16-20 mg/m2 in participants 13-18 years of age
- Group B: 250: Cetuximab 250 mg/m2 + Irinotecan 16-20 mg/m2 in participants 13-18 years of age
Arm/Group | Group A: 75 | Group A :150 | Group A: 250 | Group B: 75 | Group B: 150 | Group B: 250
Number analyzed (Participants) | 7 | 7 | 9 | 4 | 2 | 6
µg/mL | 50.5 (16.7) | 112.9 (24.7) | 163.7 (31.1) | 53.4 (21.7) | 83.1 (13.2) | 148.5 (28.1)

3. Secondary Outcome: Area Under the Curve, Extrapolated to Infinity (AUC[INF])
Description: The single dose PK of cetuximab was administered with an intravenous dose of irinotecan 16 to 20 mg/m2; AUC(INF) was evaluated based on concentration-time profile.
Time Frame: up to 168 hours after the start of the cetuximab infusion during the first 21-day cycle of the study
Measure: Geometric Mean (Standard Deviation); unit: µg•h/mL
Arm/Group | Group A: 75 | Group A :150 | Group A: 250 | Group B: 75 | Group B: 150 | Group B: 250
Number analyzed (Participants) | 7 | 7 | 9 | 4 | 2 | 6
µg•h/mL | 1598.3 (863.32) | 8871.2 (1861.1) | 17706.0 (6384.5) | 1925.2 (460.6) | 7027.3 (239.5) | 13410.4 (5484.5)

4. Secondary Outcome: Terminal Half-Life (T-Half)
Description: The single dose PK of cetuximab was administered with an intravenous dose of irinotecan 16 to 20 mg/m2; T-half was evaluated based on concentration-time profile.
Time Frame: up to 168 hours after the start of the cetuximab infusion during the first 21-day cycle of the study
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A: 75 | Group A :150 | Group A: 250 | Group B: 75 | Group B: 150 | Group B: 250
Number analyzed (Participants) | 7 | 7 | 9 | 4 | 2 | 6
hours | 31.0 (13.9) | 75.2 (18.7) | 110.3 (43.1) | 37.9 (6.3) | 61.1 (10.5) | 81.9 (20.4)

5. Secondary Outcome: Clearance Corrected for Body Surface Area (CL/BSA)
Description: The single dose PK of cetuximab was administered with an intravenous dose of irinotecan 16 to 20 mg/m2; CL/BSA was evaluated based on concentration-time profile.
Time Frame: up to 168 hours after the start of the cetuximab infusion during the first 21-day cycle of the study
Measure: Mean (Standard Deviation); unit: L/h/m2
Arm/Group | Group A: 75 | Group A :150 | Group A: 250 | Group B: 75 | Group B: 150 | Group B: 250
Number analyzed (Participants) | 7 | 7 | 9 | 4 | 2 | 6
L/h/m2 | 0.057 (0.041) | 0.017 (0.004) | 0.015 (0.005) | 0.040 (0.010) | 0.021 (0.001) | 0.020 (0.009)

6. Secondary Outcome: Volume of Distribution at Steady State Corrected for Body Surface Area (VSS/BSA)
Description: The single dose PK of cetuximab was administered with an intravenous dose of irinotecan 16 to 20 mg/m2; VSS/BSA was evaluated based on concentration-time profile.
Time Frame: up to 168 hours after the start of the cetuximab infusion during the first 21-day cycle of the study
Measure: Mean (Standard Deviation); unit: L/m2
Groups:
- Group A: 150: Cetuximab 150 mg/m2 + 16-20 mg/m2 in participants 1-12 years of age
Arm/Group | Group A: 75 | Group A: 150 | Group A: 250 | Group B: 75 | Group B: 150 | Group B: 250
Number analyzed (Participants) | 7 | 7 | 9 | 4 | 2 | 6
L/m2 | 2.081 (0.666) | 1.860 (0.564) | 2.157 (0.362) | 2.138 (0.453) | 1.887 (0.262) | 2.179 (0.250)

7. Secondary Outcome: Tumor Response
Description: Non-central nervous system (CNS) tumors evaluated using Response Evaluation Criteria In Solid Tumors (RECIST), criteria to define when cancer patients improve ("respond"), stay the same ("stable"), or worsen ("progression"). CNS tumors evaluated based on measurements by investigator, dependence on corticosteroids, and neurologic exam.
Time Frame: Every other 21-day cycle
Population: All treated subjects
Measure: Number; unit: Participants
Arm/Group | CNS Primary Tumor | Non-CNS Primary Tumor
Number analyzed (Participants) | 26 | 20
Participants
  Partial Response | 2 | 0
  Stable Disease | 10 | 8
  Progressive Disease | 10 | 11
  Not Assessable/Unable to Determine | 4 | 1

8. Secondary Outcome: Human Anti-cetuximab Antibody (HACA) Response
Description: In order to be considered positive for anti-cetuximab a sample had to: 1) be evaluable (i.e., have a pre and at least one post-treatment timepoint), 2) have an anti-cetuximab value > 7 ng/mL and 3) have a post-treatment sample at least twice the pre-treatment level.
Time Frame: Blood was drawn immediately prior to cetuximab infusions, on a 21-day cycle
Population: Cohort comprises all enrolled participants who were tested for HACA. Evaluable participants had normal baseline HACA (≤ 7 ng/dL) and ≥1 postbaseline HACA levels; unevaluable participants either did not have enough sample for analysis or did not have a pre- and postinfusion sample for immunogenicity.
Measure: Number; unit: Participants
Arm/Group | Number of Participants
Number analyzed (Participants) | 42
Participants
  Evaluable Participants | 27
  Unevaluable Participants | 15
  Participants with positive HACA level | 1

9. Secondary Outcome: Number of Deaths, Serious Adverse Events (SAEs), and Adverse Events (AEs)
Description: Toxicity assessments performed at least weekly from the 1st dose of study drug until at least 30 days after the final dose of study drug and thereafter every 4 weeks until all study-related toxicities resolved, returned to baseline, or were deemed irreversible, whichever was longer. Grade 3=severe AE; grade 4=disabling or life threatening.
Time Frame: Weekly throughout the study and every 4 weeks thereafter
Population: All treated patients
Measure: Number; unit: Participants
Arm/Group | Group A: 75/20 | Group A: 150/20 | Group A 150/16 | Group A: 250/16 | Group B: 75/20 | Group B: 150/20 | Group B: 250/20
Number analyzed (Participants) | 6 | 6 | 3 | 12 | 8 | 4 | 7
Participants
  Deaths (total) | 0 | 5 | 2 | 5 | 3 | 1 | 1
  Deaths within 30 days of last dose | 0 | 2 | 0 | 3 | 0 | 0 | 1
  SAEs | 2 | 4 | 0 | 6 | 5 | 3 | 4
  AEs leading to discontinuation of study treatment | 0 | 1 | 0 | 0 | 2 | 1 | 0
  Grade 3-4 AEs | 4 | 4 | 2 | 5 | 7 | 4 | 4

10. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RPIID) of Cetuximab in Combination With Irinotecan
Description: MTD of cetuximab intravenous (IV) weekly + irinotecan IV x5 days x2 weeks (in a 3-week cycle) and RPIID of cetuximab IV weekly, as measured by dose-limiting toxicities (see outcome measure 2)
Time Frame: Continuous assessment of safety throughout the entire study period and determination of doe-limiting toxicities during and at the end of Cycle 1.
Population: As-treated population
Measure: Number; unit: mg/m2
Arm/Group | Group A (Ages 1-12 Years) | Group B (Ages 13-18 Years)
Number analyzed (Participants) | 27 | 19
mg/m2
  MTD cetuximab (in combination w/ irinotecan) | 250 | 250
  MTD irinotecan (in combination w/ cetuximab) | 16 | 20
  RPIID cetuximab (in combination with irinotecan) | 250 | 250
  RPIID irinotecan (in combination with cetuximab) | 16 | 20

11. Secondary Outcome: Grade 3-4 Laboratory Abnormalities - Leukopenia
Description: Blood samples were collected at selected times (pretreatment visit, prior to each treatment cycle, weekly, and at the end of treatment) for clinical laboratory evaluations. Grade 3= Severe AE; Grade 4=Life-threatening or disabling AE
Time Frame: pretreatment visit, prior to each treatment cycle, weekly, and at the end of treatment
Measure: Number; unit: Participants
Groups:
- Group A 75/20: Cetuximab 75 mg/m2 + Irinotecan 20 mg/m2 in participants 1-12 years
- Group A 150/16: Cetuximab 150 mg/m2 + Irinotecan 20 mg/m2 in participants 1-12 years of age
- Group A 150/20: Cetuximab 150 mg/m2 + Irinotecan 16 mg/m2 in participants 1-12 years of age
- Group A 250/16: Cetuximab 250 mg/m2 + Irinotecan 16 mg/m2 in participants 1-12 years of age
- Group B 75/20: Cetuximab 75 mg/m2 + Irinotecan 20 mg/m2 in participants 13-18 years of age
- Group B 150/20: Cetuximab 150 mg/m2 + Irinotecan 20 mg/m2 in subjects 13-18 years of age
- Group B 250/20: Cetuximab 250 mg/m2 + Irinotecan 20 mg/m2 in participants 13-18 years of age
Arm/Group | Group A 75/20 | Group A 150/16 | Group A 150/20 | Group A 250/16 | Group B 75/20 | Group B 150/20 | Group B 250/20
Number analyzed (Participants) | 6 | 3 | 6 | 12 | 7 | 4 | 7
Participants | 3 | 0 | 3 | 4 | 2 | 2 | 4

12. Secondary Outcome: Grade 3-4 Laboratory Abnormalities - Neutropenia
Description: Blood samples were collected at selected times (pretreatment visit, prior to each treatment cycle, weekly, and at the end of treatment) for clinical laboratory evaluations. Grade 3= Severe and undesirable AE; Grade 4=Life-threatening or disabling AE
Time Frame: pretreatment visit, prior to each treatment cycle, weekly, and at the end of treatment
Measure: Number; unit: Participants
Arm/Group | Group A 75/20 | Group A 150/16 | Group A 150/20 | Group A 250/16 | Group B 75/20 | Group B 150/20 | Group B 250/20
Number analyzed (Participants) | 6 | 3 | 4 | 10 | 6 | 3 | 6
Participants | 3 | 0 | 3 | 3 | 3 | 1 | 4

13. Secondary Outcome: Grade 3-4 Laboratory Abnormalities - Thrombocytopenia
Description: Blood samples collected at selected times (pretreatment visit, prior to each treatment cycle, weekly, and at the end of treatment) for clinical laboratory evaluations. Grade 3= Severe AE; Grade 4=Life-threatening or disabling AE
Time Frame: pretreatment visit, prior to each treatment cycle, weekly, and at the end of treatment
Measure: Number; unit: Participants
Arm/Group | Group A 75/20 | Group A 150/16 | Group A 150/20 | Group A 250/16 | Group B 75/20 | Group B 150/20 | Group B 250/20
Number analyzed (Participants) | 6 | 3 | 6 | 12 | 7 | 4 | 7
Participants | 1 | 0 | 3 | 2 | 0 | 0 | 4

14. Secondary Outcome: Grade 3/4 Laboratory Abnormalities - Hypomagnesemia
Description: as for outcome 11
Time Frame: pretreatment visit, prior to each treatment cycle, weekly, and at the end of treatment
Measure: Number; unit: Participants
Arm/Group | Group A 75/20 | Group A 150/16 | Group A 150/20 | Group A 250/16 | Group B 75/20 | Group B 150/20 | Group B 250/20
Number analyzed (Participants) | 0 | 0 | 0 | 12 | 0 | 0 | 0
Participants |  |  |  | 1 |  |  |

ADVERSE EVENTS:
Arm/Group | 01 75 mg/m2 CET + 20 mg/m2 IRI | 02 150 mg/m2 CET + 20 mg/m2 IRI | 03 150 mg/m2 CET + 16 mg/m2 IRI | 04 250 mg/m2 CET + 16 mg/m2 IRI | 05 250 mg/m2 CET + 20 mg/m2 IRI
Serious Adverse Events (participants affected / at risk) | 7/14 | 7/10 | 0/3 | 6/12 | 4/7
Other Adverse Events (participants affected / at risk) | 14/14 | 8/10 | 3/3 | 12/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 01 75 mg/m2 CET + 20 mg/m2 IRI (N=14) | 02 150 mg/m2 CET + 20 mg/m2 IRI (N=10) | 03 150 mg/m2 CET + 16 mg/m2 IRI (N=3) | 04 250 mg/m2 CET + 16 mg/m2 IRI (N=12) | 05 250 mg/m2 CET + 20 mg/m2 IRI (N=7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
NEUTROPHIL COUNT (Investigations) | 0 | 0 | 0 | 0 | 1
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
CRANIAL NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
DISEASE PROGRESSION (General disorders) | 0 | 1 | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
HAEMOGLOBIN (Investigations) | 0 | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 3
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
WHITE BLOOD CELL COUNT (Investigations) | 0 | 0 | 0 | 0 | 1
CATHETER RELATED INFECTION (Infections and infestations) | 1 | 1 | 0 | 0 | 0
CENTRAL LINE INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ELECTIVE SURGERY (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
ILEUS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
INFUSION RELATED REACTION (General disorders) | 0 | 0 | 0 | 1 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 2 | 1 | 0 | 0 | 0
PYREXIA (General disorders) | 2 | 3 | 0 | 1 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 1 | 0 | 2 | 0
GRANULOCYTE COUNT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 1
PAIN (General disorders) | 1 | 0 | 0 | 0 | 0
PLATELET COUNT (Investigations) | 0 | 0 | 0 | 0 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 1
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 2 | 1 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
ROTAVIRUS INFECTION (Infections and infestations) | 1 | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
FAECAL INCONTINENCE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
FATIGUE (General disorders) | 2 | 0 | 0 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
BLOOD BICARBONATE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 1
GALLBLADDER OBSTRUCTION (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
HYDROCEPHALUS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 1 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
CHILLS (General disorders) | 0 | 2 | 0 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
LETHARGY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
NECROSIS (General disorders) | 1 | 0 | 0 | 0 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
SPEECH DISORDER (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 01 75 mg/m2 CET + 20 mg/m2 IRI (N=14) | 02 150 mg/m2 CET + 20 mg/m2 IRI (N=10) | 03 150 mg/m2 CET + 16 mg/m2 IRI (N=3) | 04 250 mg/m2 CET + 16 mg/m2 IRI (N=12) | 05 250 mg/m2 CET + 20 mg/m2 IRI (N=7)
ADVERSE EVENT (General disorders) | 1 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE (Investigations) | 1 | 0 | 0 | 1 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BLOOD BILIRUBIN (Investigations) | 0 | 0 | 0 | 1 | 0
CHAPPED LIPS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 3 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 7 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
EAR LOBE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
FLUSHING (Vascular disorders) | 1 | 0 | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 3 | 0 | 1 | 0 | 1
HAIR GROWTH ABNORMAL (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
INJECTION SITE REACTION (General disorders) | 1 | 0 | 0 | 0 | 0
LOCALISED OEDEMA (General disorders) | 0 | 0 | 0 | 1 | 0
MELAENA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 1 | 0 | 1 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 1
NEUTROPHIL COUNT (Investigations) | 1 | 0 | 0 | 0 | 1
NEUTROPHIL COUNT INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
WEIGHT INCREASED (Investigations) | 2 | 0 | 1 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
ASPARTATE AMINOTRANSFERASE (Investigations) | 2 | 0 | 0 | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 0 | 1 | 0 | 0 | 0
BLOOD UREA DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
CARBON DIOXIDE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 0 | 1 | 0
CRANIAL NEUROPATHY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
HAEMOGLOBIN (Investigations) | 1 | 0 | 0 | 1 | 0
HAEMOGLOBIN ABNORMAL (Investigations) | 0 | 0 | 1 | 0 | 0
HALLUCINATION (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
HANGNAIL (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 9 | 4 | 2 | 7 | 4
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
MOOD ALTERED (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
PHARYNGEAL ERYTHEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 5 | 5
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 1 | 1
WHITE BLOOD CELL COUNT (Investigations) | 1 | 0 | 0 | 0 | 1
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 0 | 1 | 0 | 0
CENTRAL LINE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 2 | 0 | 0 | 1 | 2
DEPRESSED MOOD (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
ENURESIS (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
EYELASH THICKENING (Eye disorders) | 0 | 0 | 0 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
INFUSION RELATED REACTION (General disorders) | 1 | 0 | 0 | 0 | 0
LIP ULCERATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
LYMPHOCYTE COUNT (Investigations) | 1 | 0 | 0 | 0 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0 | 1
PROCTALGIA (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
PROTEIN TOTAL INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 5 | 3 | 0 | 4 | 2
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 0
STRABISMUS (Eye disorders) | 1 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 2 | 0 | 1 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
ACNE (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
ANURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 0 | 1
BLOOD SODIUM DECREASED (Investigations) | 2 | 0 | 0 | 0 | 0
CATHETER SITE INFECTION (Infections and infestations) | 1 | 0 | 0 | 1 | 0
CERUMEN IMPACTION (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 3 | 1 | 1 | 5 | 1
CULTURE STOOL POSITIVE (Investigations) | 1 | 0 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 2
EYE DISORDER (Eye disorders) | 0 | 0 | 0 | 2 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
GRANULOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
INFUSION SITE PAIN (General disorders) | 0 | 1 | 0 | 0 | 0
LOWER EXTREMITY MASS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 11 | 5 | 0 | 7 | 6
NEUTROPHIL COUNT DECREASED (Investigations) | 2 | 0 | 0 | 0 | 1
PAIN (General disorders) | 2 | 0 | 0 | 1 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PLATELET COUNT (Investigations) | 0 | 0 | 0 | 1 | 1
PSYCHIATRIC SYMPTOM (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 11 | 5 | 1 | 9 | 6
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1
ARTHROPOD STING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
BLOOD CHLORIDE DECREASED (Investigations) | 2 | 0 | 0 | 0 | 0
BLOOD CHLORIDE INCREASED (Investigations) | 2 | 0 | 0 | 0 | 0
BLOOD MAGNESIUM DECREASED (Investigations) | 2 | 0 | 0 | 0 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BLOOD URIC ACID DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
DEAFNESS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 0
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 0 | 1 | 0
GLYCOSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
HIRSUTISM (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
HYPERCHLORHYDRIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 1 | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 3 | 1 | 0 | 1 | 1
LOCALISED INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1
MALAISE (General disorders) | 1 | 0 | 0 | 1 | 0
MUCOUS STOOLS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 2 | 0
PROTEIN TOTAL DECREASED (Investigations) | 1 | 0 | 1 | 0 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
TONGUE ULCERATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 5 | 1 | 9 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 0 | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1
BLOOD AMYLASE DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BLOOD CALCIUM DECREASED (Investigations) | 1 | 0 | 1 | 0 | 0
CROUP INFECTIOUS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
ENCEPHALITIS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
EXOPHTHALMOS (Eye disorders) | 0 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 4 | 4 | 1 | 4 | 1
FLATULENCE (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
IRRITABILITY (General disorders) | 0 | 1 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
PAINFUL DEFAECATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 2 | 0 | 0 | 1 | 1
SKIN INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 | 2 | 0 | 1 | 0
ANOREXIA (Metabolism and nutrition disorders) | 6 | 3 | 0 | 6 | 2
ANXIETY (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
ASTHENIA (General disorders) | 1 | 1 | 0 | 0 | 0
BLOOD BICARBONATE DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
BLOOD POTASSIUM ABNORMAL (Investigations) | 0 | 0 | 1 | 0 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 2 | 0 | 1 | 0 | 1
BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CATHETER SITE PAIN (General disorders) | 1 | 0 | 0 | 1 | 0
CATHETER SITE RASH (General disorders) | 0 | 0 | 0 | 1 | 0
CONJUNCTIVITIS INFECTIVE (Infections and infestations) | 1 | 0 | 0 | 0 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 11 | 7 | 2 | 10 | 6
DIZZINESS (Nervous system disorders) | 2 | 1 | 0 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
EMOTIONAL DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
HAEMOLYSIS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
HYDROCEPHALUS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 0 | 1 | 0 | 0 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
INTERNATIONAL NORMALISED RATIO (Investigations) | 1 | 0 | 0 | 0 | 0
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 | 0 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1 | 1 | 0
PHOTOPHOBIA (Eye disorders) | 1 | 0 | 0 | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 1 | 0 | 1
POLYURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
SKIN INDURATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
TREMOR (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 0 | 1 | 1 | 0
VIRUS CULTURE POSITIVE (Investigations) | 1 | 0 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 4 | 4 | 1 | 8 | 2
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
BLOOD ALBUMIN (Investigations) | 0 | 0 | 0 | 0 | 1
BLOOD ALBUMIN DECREASED (Investigations) | 2 | 0 | 1 | 0 | 0
BLOOD CULTURE POSITIVE (Investigations) | 0 | 0 | 0 | 1 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 3 | 0 | 0 | 0 | 0
CATHETER RELATED COMPLICATION (General disorders) | 0 | 0 | 1 | 0 | 0
CHILLS (General disorders) | 0 | 0 | 1 | 2 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 1 | 1 | 1
CONVULSION (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 3 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
GROWTH OF EYELASHES (Eye disorders) | 3 | 0 | 0 | 0 | 0
INFUSION SITE EXTRAVASATION (General disorders) | 0 | 0 | 0 | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
NAIL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 3 | 0
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
PARONYCHIA (Infections and infestations) | 2 | 1 | 0 | 0 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 1
SKIN CANDIDA (Infections and infestations) | 0 | 1 | 0 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
SPEECH DISORDER (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 3 | 2 | 0 | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.